CLINICAL TRIAL: NCT00925600
Title: A Double-blind, Placebo-controlled Study to Evaluate New or Worsening Lens Opacifications in Subjects With Non-metastatic Prostate Cancer Receiving Denosumab for Bone Loss Due to Androgen-Deprivation Therapy
Brief Title: Evaluation of New or Worsening Lens Opacifications in Men With Non-metastatic Prostate Cancer Receiving Denosumab for Bone Loss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20080560; 2009-012076-26 (EudraCT Number)
Record Dates: First submitted 2009-06-18; First posted 2009-06-22 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Cancer; Cataract; Low Bone Mineral Density; Osteopenia; Osteoporosis; Prostate Cancer
Keywords: Lens Opacification; Bone Loss; Androgen Deprivation Therapy; Non-metastatic prostate cancer
MeSH Terms: conditions — Neoplasms; Cataract; Bone Diseases, Metabolic; Osteoporosis; Prostatic Neoplasms | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo administered by subcutaneous injection on Day 1 and at Month 6.
  Interventions: Biological: Placebo
- Denosumab (Experimental): Participants received denosumab 60 mg administered by subcutaneous injection on Day 1 and at Month 6.
  Interventions: Biological: Denosumab

INTERVENTIONS:
Biological: Denosumab — Prefilled syringe for subcutaneous (SC) injection administered at a dose of 60 mg
  Other Names: Prolia®
  Arms: Denosumab
Biological: Placebo — Prefilled syringe for subcutaneous (SC) injection
  Arms: Placebo

SUMMARY:
This is a phase 3, randomized, double-blind, placebo-controlled study to evaluate new or worsening lens opacifications in men with non-metastatic prostate cancer receiving denosumab for bone loss due to androgen deprivation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥ 30 years of age with non-metastatic prostate cancer, having undergone bilateral orchiectomy or initiated androgen deprivation therapy (ADT) with gonadotropin-releasing hormone (GnRH) agonists and is expected to continue on ADT for at least 12 months
* Adequate visual accuracy allowing eye testing
* Bone Mineral Density (BMD) requirements: Osteopenia if under 70 years of age; Osteopenia or normal BMD if over 70 years of age
* Signed informed consent

Exclusion Criteria:

* Previous surgery for cataracts in both eyes, current diagnosis of cataracts, cataracts surgery foreseen in the near future, or ocular disease leading to visual loss
* Diagnosis of osteoporosis

Ages: 30 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 769 (Actual)
Dates: Start 2009-11-30 (Actual); Primary Completion 2016-05-12 (Actual); Study Completion 2016-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (148):
- United States (48):
  - Research Site, Anaheim, California
  - Research Site, Laguna Hills, California
  - Research Site, Murrieta, California
  - Research Site, San Diego, California
  - Research Site, San Luis Obispo, California
  - Research Site, Denver, Colorado
  - Research Site, Englewood, Colorado
  - Research Site, Middlebury, Connecticut
  - Research Site, New Britain, Connecticut
  - Research Site, Trinity, Florida
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Greenwood, Indiana
  - Research Site, West Des Moines, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Shreveport, Louisiana
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Greenbelt, Maryland
  - Research Site, Grand Rapids, Michigan
  - Research Site, Sartell, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Berlin, New Jersey
  - Research Site, Brick, New Jersey
  - Research Site, Englewood, New Jersey
  - Research Site, Lawrenceville, New Jersey
  - Research Site, Mount Laurel, New Jersey
  - Research Site, Albany, New York
  - Research Site, Garden City, New York
  - Research Site, Kingston, New York
  - Research Site, New York, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Syracuse, New York
  - Research Site, Gastonia, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Bala-Cynwyd, Pennsylvania
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Temple, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Salem, Virginia
- Australia (4):
  - Research Site, Wahroonga, New South Wales
  - Research Site, Herston, Queensland
  - Research Site, Bentleigh East, Victoria
  - Research Site, Ringwood East, Victoria
- Bulgaria (3):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (19):
  - Research Site, Kelowna, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Barrie, Ontario
  - Research Site, Brampton, Ontario
  - Research Site, Brantford, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Guelph, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, North Bay, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
- Czechia (11):
  - Research Site, Benešov
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Jindřichův Hradec
  - Research Site, Kroměříž
  - Research Site, Nový Jičín
  - Research Site, Olomouc
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Ústí nad Labem
  - Research Site, Zlín
- France (2):
  - Research Site, Lyon Cédex 3
  - Research Site, Paris
- Greece (6):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Larissa
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hungary (6):
  - Research Site, Baja
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Szeged
- India (7):
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Bangalore, Karnataka
  - Research Site, Aurangabad, Maharashtra
  - Research Site, Nashik, Maharashtra
  - Research Site, Ludhiana, Punjab
  - Research Site, Madurai, Tamil Nadu
  - Research Site, Kolkata, West Bengal
- Latvia (2):
  - Research Site, Jelgava
  - Research Site, Riga
- Research Site, Distrito Federal, Mexico
- New Zealand (4):
  - Research Site, Christchurch
  - Research Site, Takapuna, North Shore City
  - Research Site, Tauranga
  - Research Site, Whangarei
- Poland (12):
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Katowice
  - Research Site, Mysłowice
  - Research Site, Opole
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Siedlce
  - Research Site, Szczecin
  - Research Site, Słupsk
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (4):
  - Research Site, Ivanovo
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Rostov-on-Don
- Slovakia (5):
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Martin
  - Research Site, Nitra
  - Research Site, Trenčín
- Slovenia (3):
  - Research Site, Celje
  - Research Site, Ljubljana
  - Research Site, Slovenj Gradec
- South Africa (5):
  - Research Site, Paarl, Western Cape
  - Research Site, George
  - Research Site, Kempton Park
  - Research Site, Port Elizabeth
  - Research Site, Tygerberg
- Ukraine (6):
  - Research Site, Chernivtsi
  - Research Site, Dnipropetrovsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Uzhhorod
  - Research Site, Zaporizhzhya

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 125 centers in 18 countries: Australia, Bulgaria, Canada, the Czech Republic, France, Greece, Hungary, India, Latvia, Mexico, New Zealand, Poland, Russia, Slovakia, Slovenia, South Africa, Ukraine, and the United States.
  The first participant enrolled on 30 November 2009 and the last participant enrolled on 04 May 2015.
Pre-assignment Details: Participants were randomly assigned to receive denosumab or placebo in a 1:1 allocation ratio. Randomization was stratified on the basis of screening Lens Opacities Classification System (LOCS) III status (< 3.0 at all sites versus ≥ 3.0 at any site); age group (< 75, ≥ 75 years), and patient-reported history of cataract (yes/no).
Groups:
- Placebo: Participants randomized to receive placebo administered by subcutaneous injection on Day 1 and at Month 6.
- Denosumab: Participants randomized to receive denosumab 60 mg administered by subcutaneous injection on Day 1 and at Month 6.
Period: Overall Study
Arm/Group | Placebo | Denosumab
Started | 386 | 383
Received Treatment | 383 (Three participants received at least 1 dose of denosumab in error) | 382
Completed | 354 | 355
Not Completed | 32 | 28
Not completed — Withdrawal by Subject | 16 | 14
Not completed — Death | 4 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Disease Progression | 1 | 3
Not completed — Administrative Decision | 1 | 1
Not completed — Noncompliance | 2 | 0
Not completed — Ineligibility Determined | 2 | 0
Not completed — Protocol Deviation | 0 | 1
Not completed — Requirement for Alternative Therapy | 0 | 1
Not completed — Other | 3 | 1
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Denosumab | Total
Number analyzed (Participants) | 386 | 383 | 769
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (7.0) | 71.1 (7.2) | 71.0 (7.1)
Age, Customized [Number; unit: participants]
  18 - 64 years | 73 | 66 | 139
  65 - 74 years | 189 | 194 | 383
  75 - 84 years | 119 | 116 | 235
  ≥ 85 years | 5 | 7 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 386 | 383 | 769
Race/Ethnicity, Customized [Number; unit: participants]
  White | 359 | 346 | 705
  Black (or African American) | 12 | 11 | 23
  Hispanic/Latino | 1 | 9 | 10
  Other | 7 | 8 | 15
  Asian | 7 | 7 | 14
  Japanese | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
Presence of Cataract(s) [Number; unit: participants] — From baseline medical history
  participants
    Yes | 59 | 63 | 122
    No | 327 | 320 | 647
Presence of Diabetes [Number; unit: participants] — From baseline medical history
  participants
    Yes | 70 | 61 | 131
    No | 316 | 322 | 638
Received Androgen-deprivation Therapy (ADT) [Number; unit: participants]
  Yes | 350 | 353 | 703
  No | 36 | 30 | 66
Orchiectomy (Surgical Castration) [Number; unit: participants]
  Yes | 58 | 51 | 109
  No | 328 | 332 | 660
Screening Lens Opacities Classification System (LOCS) III Status [Number; unit: participants] — The Lens Opacities Classification System III (LOCS III) is a slit lamp based opacification grading method. Photographs of slit lamp cross-sections of the lens are used as references for grading nuclear opalescence (NO) and nuclear color (NC), and photographs of the lens seen by retroillumination are used as references for grading cortical (C) and posterior subcapsular (P) cataract. Opacification severity is graded on a decimal scale, scores can range from 0.1 to 6.9 for NO and NC and from 0.1 to 5.9 for C and P. For each opacification type the higher grading scores indicate greater severity.
  participants
    < 3.0 at all sites [P, C, and NO] | 299 | 299 | 598
    ≥ 3.0 at any of these sites | 87 | 84 | 171
Participant-reported History of Cataract [Number; unit: participants] — Participant-reported history of cataracts was a study stratification factor.
  participants
    Yes | 35 | 35 | 70
    No | 351 | 348 | 699

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Lens Opacification Event Development or Progression by Month 12
Description: The Lens Opacities Classification System III (LOCS III) is a slit lamp based opacification grading method. Photographs of slit lamp cross-sections of the lens are used as references for grading nuclear opalescence (NO) and nuclear color (NC), and photographs of the lens seen by retroillumination are used as references for grading cortical (C) and posterior subcapsular (P) cataract. Opacification severity is graded on a decimal scale, scores can range from 0.1 to 6.9 for NO and NC and from 0.1 to 5.9 for C and P. For each opacification type the higher grading scores indicate greater severity. Lens opacification event development or progression by month 12 was based on a change of ≥ 1.0 in P, ≥ 1.0 in C, or ≥ 0.7 in NO in the LOCS III score from baseline.
Time Frame: 12 months
Population: The lens opacification analysis set includes randomized participants who received ≥1 dose of study drug, had an evaluable baseline and at least 1 evaluable post-baseline LOCS III assessment at the corresponding lens site. Three participants randomized to placebo who received ≥ 1 dose of denosumab in error are analyzed in the denosumab group.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 374 | 379
percentage of participants | 33.2 | 33.5
Statistical Analysis 1: Comparison: Placebo vs Denosumab; The primary endpoint was summarized with the point estimate of absolute risk difference (difference in incidence rates, denosumab minus placebo) and the corresponding 95% confidence interval using the Mantel-Haenszel method adjusting for the stratification factors: baseline LOCS III status (< 3.0 at all sites [P, C, and NO] vs. ≥ 3.0 at any of these sites), age group (< 75, ≥ 75 years), and patient-reported history of cataract (yes/no); Test type: Non-Inferiority or Equivalence — Non-inferiority was demonstrated if the upper bound of the 97.5% one-sided confidence interval, or equivalently upper bound of two-sided 95% confidence interval was less than the pre-specified non-inferiority bound of 10%; p = 0.0026, Mantel Haenszel; Risk Difference (RD) = 0.4, 95% CI 2-sided [-6.3 to 7.2], Standard Error of Mean 3.4

2. Other Pre Specified Outcome: Percentage of Participant With Lens Opacification Event Development or Progression by Month 12 Based on a Change of ≥ 1.5 in P, ≥ 1.5 in C, or ≥ 1.5 in NO in the LOCS III Score
Description: The Lens Opacities Classification System III (LOCS III) is a slit lamp based opacification grading method. Photographs of slit lamp cross-sections of the lens are used as references for grading nuclear opalescence (NO) and nuclear color (NC), and photographs of the lens seen by retroillumination are used as references for grading cortical (C) and posterior subcapsular (P) cataract. Opacification severity is graded on a decimal scale, scores can range from 0.1 to 6.9 for NO and NC and from 0.1 to 5.9 for C and P. For each opacification type the higher grading scores indicate greater severity. Lens opacification event development or progression by month 12 was based on a change ≥ 1.5 in P, ≥ 1.5 in C, or ≥ 1.5 in NO in the LOCS III score from baseline.
Time Frame: 12 months
Population: The lens opacification analysis set includes randomized participants who received ≥1 dose of study drug, had an evaluable baseline and at least 1 evaluable post-baseline LOCS III assessment at the corresponding lens site. Three participants randomized to placebo who eceived ≥ 1 dose of denosumab in error are analyzed in the denosumab group.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 374 | 379
percentage of participants | 10.7 | 8.4
Statistical Analysis 1: Comparison: Placebo vs Denosumab; The point estimate of absolute risk difference (difference in incidence rates, denosumab minus placebo) and the corresponding 95% confidence interval was constructed using the Mantel-Haenszel method adjusting for the stratification factors: baseline LOCS III status (< 3.0 at all sites [P, C, and NO] vs. ≥ 3.0 at any of these sites), age group (< 75, ≥ 75 years), and patient-reported history of cataract (yes/no); Test type: Superiority or Other; Risk Difference (RD) = -2.2, 95% CI 2-sided [-6.4 to 2.0], Standard Error of Mean 2.1

3. Other Pre Specified Outcome: Percentage of Participants With Lens Opacification Event Development or Progression by Month 6
Description: The Lens Opacities Classification System III (LOCS III) is a slit lamp based opacification grading method. Photographs of slit lamp cross-sections of the lens are used as references for grading nuclear opalescence (NO) and nuclear color (NC), and photographs of the lens seen by retroillumination are used as references for grading cortical (C) and posterior subcapsular (P) cataract. Opacification severity is graded on a decimal scale, scores can range from 0.1 to 6.9 for NO and NC and from 0.1 to 5.9 for C and P. For each opacification type the higher grading scores indicate greater severity. Lens opacification event development or progression by month 6 was based on a change of ≥ 1.0 in P, ≥ 1.0 in C, or ≥ 0.7 in NO in the LOCS III score from baseline.
Time Frame: 6 months
Population: Lens opacification analysis set includes randomized participants who received ≥1 dose of study drug, had an evaluable baseline and at least 1 evaluable post-baseline LOCS III assessment at the corresponding lens site at or before month 6. Three participants randomized to placebo who received denosumab in error are analyzed in the denosumab group.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 374 | 379
percentage of participants | 19.3 | 19.0
Statistical Analysis 1: Comparison: Placebo vs Denosumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Risk Difference (RD) = -0.3, 95% CI 2-sided [-5.9 to 5.3], Standard Error of Mean 2.9

4. Other Pre Specified Outcome: Percentage of Participants With Confirmed Lens Opacification Event Development or Progression by Month 12
Description: The Lens Opacities Classification System III (LOCS III) is a slit lamp based opacification grading method. Photographs of slit lamp cross-sections of the lens are used as references for grading nuclear opalescence (NO) and nuclear color (NC), and photographs of the lens seen by retroillumination are used as references for grading cortical (C) and posterior subcapsular (P) cataract. Opacification severity is graded on a decimal scale, scores can range from 0.1 to 6.9 for NO and NC and from 0.1 to 5.9 for C and P. For each opacification type the higher grading scores indicate greater severity.
  Lens opacification event development or progression by month 12 was based on a change of ≥ 1.0 in P, ≥ 1.0 in C, or ≥ 0.7 in NO in the LOCS III score from baseline. A confirmed lens opacification event development or progression was defined as 2 directly subsequent events per protocol assessments at the same location (P, C, NO) using LOCS III as above.
Time Frame: 12 months
Population: Lens opacification analysis set with at least two post-baseline LOCS III measurements by month 12.
  Three participants randomized to placebo who received at least 1 dose of denosumab in error are analyzed in the denosumab group.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 361 | 367
percentage of participants | 18.3 | 16.1
Statistical Analysis 1: Comparison: Placebo vs Denosumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Risk Difference (RD) = -2.2, 95% CI 2-sided [-7.6 to 3.3], Standard Error of Mean 2.8

5. Other Pre Specified Outcome: Percentage of Participants With a Decrease From Baseline in Best Corrected Visual Acuity (BCVA) of ≥ 10 Letters
Description: The best corrected visual acuity (BCVA) is the best vision one can achieve with correction (such as eye glasses) as measured on an eye chart. BCVA was assessed by a trained ophthalmologist using the Early Treatment Diabetic Retinopathy Study (ETDRS) eye chart at 4 meters. The modified University of Crete ETDRS chart was used in Ukraine, Greece, Russia and Bulgaria, which do not use the Roman alphabet. The 2000 series revised ETDRS chart was used to assess the change in all other countries.
  The letter score was calculated based on the number of letters that were correctly identified; higher letter scores correspond to better visual acuity.
Time Frame: Baseline and Months 3, 6, 9 and 12
Population: Lens opacification analysis set with evaluable assessments at both baseline and the time point of interest in the same eye (as indicated by "n"). Three participants randomized to placebo who received at least 1 dose of denosumab in error are analyzed in the denosumab group.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 374 | 379
percentage of participants
  Month 3 (n = 372, 375) | 5.4 | 6.1
  Month 6 (n = 355, 357) | 4.2 | 6.4
  Month 9 (n = 350, 346) | 4.6 | 6.6
  Month 12 (n = 343, 342) | 5.2 | 7.3

6. Other Pre Specified Outcome: Change From Baseline in Refraction Needed to Achieve BCVA
Description: Refraction error was measured using a phoropter. The change from baseline in spherical refraction error needed to achieve BCVA is reported.
Time Frame: Baseline and months 3, 6, 9, and 12
Population: Lens opacification analysis set with evaluable assessments at both baseline and each time point in the same eye.
  n=the number of evaluable eyes in the lens opacification analysis set at the corresponding time point; 3 participants randomized to placebo who received denosumab in error are analyzed in the denosumab group.
Measure: Mean (Standard Deviation); unit: diopters
Units Other Than Participants: eyes
Groups:
- Placebo - Left Eye; Placebo - Right Eye: Participants received placebo subcutaneous injection on Day 1 and at Month 6.
- Denosumab - Right Eye: Participants received denosumab 60 mg administered by subcutaneous injection on Day 1 and at Month 6.
Arm/Group | Placebo - Left Eye | Placebo - Right Eye | Denosumab | Denosumab - Right Eye
Number analyzed (Participants) | 374 | 374 | 379 | 379
Number analyzed (eyes) | 374 | 374 | 379 | 379
diopters
  Month 3 (n = 362, 358, 358, 359) | 0.01 (0.60) | 0.01 (0.49) | 0.05 (0.73) | 0.04 (0.51)
  Month 6 (n = 347, 343, 341, 344) | -0.01 (0.80) | 0.06 (0.70) | 0.06 (0.90) | 0.04 (0.59)
  Month 9 (n = 341, 339, 332, 332) | 0.00 (0.84) | 0.01 (0.73) | 0.04 (0.75) | 0.01 (0.62)
  Month 12 (n = 336, 334, 328, 329) | -0.03 (0.70) | -0.04 (0.59) | 0.03 (0.77) | 0.00 (0.48)

7. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) were assessed for severity by the investigator according to the Common Terminology Criteria for Adverse Events (CTCAE) severity grading scale, version 3.0, where Grade 1 = Mild AE, Grade 2 = Moderate AE, Grade 3 = Severe AE, Grade 4 =Life-threatening AE and Grade 5 = Death due to AE.
  Treatment-related AEs (TRAEs) include only events for which the investigator indicated there was a reasonable possibility they may have been caused by the study drug.
Time Frame: 12 months
Population: All enrolled participants who received at least one dose of study drug. Three participants randomized to the placebo group who received at least 1 dose of denosumab in error are analyzed in the denosumab group for safety.
Measure: Number; unit: participants
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 380 | 385
participants
  Any adverse event | 193 | 191
  Serious adverse events | 52 | 42
  AE leading to discontinuation of study drug | 5 | 7
  AE leading to discontinuation from study | 2 | 4
  Fatal adverse events | 4 | 3
  AE grade 3, 4, or 5 | 53 | 46
  Treatment-related adverse events | 19 | 21
  Serious treatment-related adverse events | 1 | 2
  TRAE leading to discontinuation of study drug | 1 | 3
  TRAE leading to discontinuation from study | 0 | 1
  Fatal treatment-related adverse events | 0 | 0
  TRAE grade 3, 4, or 5 | 2 | 2

ADVERSE EVENTS:
Time Frame: 12 months
Description: All enrolled participants who received at least one dose of study drug. Three participants randomized to the placebo group received at least 1 dose of denosumab in error, and are included in the denosumab group for safety.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Denosumab
Serious Adverse Events (participants affected / at risk) | 52/380 | 42/385
Other Adverse Events (participants affected / at risk) | 107/380 | 121/385
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=380) | Denosumab (N=385)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiac fibrillation (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 1
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 3
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Optic nerve disorder (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Small intestinal stenosis (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Cyst (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 0
Pseudoangina (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 1
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Radiation proctitis (Injury, poisoning and procedural complications) | 0 | 1
Urethral stricture postoperative (Injury, poisoning and procedural complications) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Connective tissue inflammation (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 4 | 1
Dementia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Encephalomalacia (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Device dislocation (Product Issues) | 0 | 1
Device malfunction (Product Issues) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=380) | Denosumab (N=385)
Anaemia (Blood and lymphatic system disorders) | 4 | 2
Atrial fibrillation (Cardiac disorders) | 3 | 4
Vertigo (Ear and labyrinth disorders) | 0 | 6
Vision blurred (Eye disorders) | 2 | 5
Constipation (Gastrointestinal disorders) | 16 | 8
Diarrhoea (Gastrointestinal disorders) | 6 | 2
Fatigue (General disorders) | 2 | 6
Oedema peripheral (General disorders) | 1 | 7
Bronchitis (Infections and infestations) | 4 | 6
Nasopharyngitis (Infections and infestations) | 7 | 10
Sinusitis (Infections and infestations) | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 6 | 5
Urinary tract infection (Infections and infestations) | 5 | 5
Chest injury (Injury, poisoning and procedural complications) | 4 | 0
Prostatic specific antigen increased (Investigations) | 0 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 5
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 6
Dizziness (Nervous system disorders) | 4 | 6
Headache (Nervous system disorders) | 3 | 6
Insomnia (Psychiatric disorders) | 3 | 6
Dysuria (Renal and urinary disorders) | 4 | 5
Haematuria (Renal and urinary disorders) | 4 | 3
Pollakiuria (Renal and urinary disorders) | 6 | 7
Urinary incontinence (Renal and urinary disorders) | 4 | 1
Urinary retention (Renal and urinary disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Hot flush (Vascular disorders) | 7 | 7
Hypertension (Vascular disorders) | 16 | 8
Hypotension (Vascular disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.